CLINICAL TRIAL: NCT03987828
Title: Long-term Outcomes After Noncurative Endoscopic Resection of Colorectal Adenocarcinoma
Brief Title: Noncurative Endoscopic Resection of Colorectal Adenocarcinoma
Acronym: NoncurativeESD
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: Non_curativeESD
Record Dates: First submitted 2019-06-11; First posted 2019-06-17 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Noncurative Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with noncurative resection after ESD for CRC were considered for additional surgical treatment. Then, they either underwent surgery with curative intent or did not, according to patients choice and surgeons indication / contraindication.

We performed a retrospective revision of outcome data by clinical report review or phone calls.

DETAILED DESCRIPTION:
Patients with noncurative resection after ESD for CRC were considered for additional surgical treatment. Then, they either underwent surgery with curative intent or did not, according to patients choice and surgeons indication / contraindication.

We performed a retrospective revision of outcome data by clinical report review or phone calls.

ELIGIBILITY:
Inclusion Criteria:

- undergoing non-curative colorectal endoscopic submucosal dissection (ESD).

Exclusion Criteria:

* Histology other than cancer (adenocarcinoma).
* History of inflammatory bowel disease (IBD).
* Genetic conditions predisposing to CR.
* Lost to follow up or less than 6 months of follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent a non-curative colorectal endoscopic submucosal dissection (ESD). Curative resection was defined as follows: en bloc resection (tumor removal in one piece without fragmentation) and R0 resection (negative horizontal and vertical resected margins) of a neoplastic (adenocarcinoma) lesion with no lymphovascular infiltration (LVI), no budding, no undifferentiated tumor (G3), no deep invasion (T1 sm3 or deeper).
  Patients are required to meet none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Survival | 6 Months
  Overall survival cancer-specific survival and disease-free survival rate after noncurative ESD.

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

REFERENCES:
- [Derived] Spadaccini M, Bourke MJ, Maselli R, Pioche M, Bhandari P, Jacques J, Haji A, Yang D, Albeniz E, Kaminski MF, Messmann H, Herreros de Tejada A, Sferrazza S, Pekarek B, Rivory J, Geyl S, Gulati S, Draganov P, Shahidi N, Hossain E, Fleischmann C, Vespa E, Iannone A, Alkandari A, Hassan C, Repici A; ESD Western Alliance (EWA). Clinical outcome of non-curative endoscopic submucosal dissection for early colorectal cancer. Gut. 2022 Sep 7;71(10):1998-2004. doi: 10.1136/gutjnl-2020-323897. PMID 35058275